CLINICAL TRIAL: NCT01370564
Title: Feasibility of an Integrated Patient Care (IPC) System Using Daily Filling Pressures
Acronym: IPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPC
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac filling pressure
MeSH Terms: conditions — Heart Failure | interventions — Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily diuretic adjustment (Other): Daily adjustments of diuretics and associated supplements based on cardiac filling pressures.
  Interventions: Drug: Diuretics

INTERVENTIONS:
Drug: Diuretics — Daily adjustments of diuretics and associated supplements based on cardiac filling pressures.

SUMMARY:
This chronic, prospective, non-randomized feasibility study is designed to evaluate the Integrated Patient Care (IPC) concept in subjects who already have either a Medtronic Chronicle Implantable Hemodynamic Monitor (IHM) or Chronicle Implantable Cardioverter Defibrillator (ICD) device implanted, and are currently enrolled in the Chronicle Offers Management to Patients with Advanced Signs & Symptoms of Heart Failure (COMPASS-HF) Extension Phase Study (IDE # G020304). The purpose of the study is to use daily cardiac filling pressures from the Chronicle device to provide timely medication adjustments (diuretics) to subjects.

DETAILED DESCRIPTION:
Subjects will be asked to transmit to the CareLink Network daily. Data specific to this study (subject's daily estimated Pulmonary Arterial Diastolic (ePAD) pressure values) will be extracted from the CareLink database and transferred to the IPC clinician website.

As each subject is enrolled, clinicians at each participating site will determine the appropriate target pressure range for each subject based on a review of the subject's pressure data. Each day after enrollment, the subject's current pressure data will be compared to a target pressure range that the clinician sets for that subject.

The patient instruction set (PtIS) is limited to a daily diuretic prescription and associated supplements, per physician discretion. The PtIS should not include adjustments of non-heart failure medications and should not include heart failure medications that are not indicated for day-to-day adjustments (e.g. ACE-Inhibitors, Angiotensin Receptor Blockers (ARBs), and Beta-Blockers). The PtIS will be sent from the IPC clinician website to the subject through a Patient Home Monitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a Chronicle IHM device (Model 9520, Model 9520B) or Chronicle ICD device (Model 7286)
* Patients who have been prescribed daily diuretic therapy for the management of heart failure
* Patients currently participating in the COMPASS-HF Extension Phase Study (IDE #G020304)
* Patients willing and able to give informed consent

Exclusion Criteria:

* Patients with non-physiologic Right Ventricular (RV) pressure values
* Patients who have diuretic resistance
* Patients who have an estimated Glomerular Filtration Rate(eGFR) <30 ml/min (recorded within the last six months)
* Patients who have a Chronicle IHM device (Model 9520) that was implanted as part of the Pulmonary Arterial Hypertension (PAH) Pilot Study (IDE #G020303)
* Patients who do not have the ability to actively participate in the management of their own heart failure care (determine by physician discretion)(e.g. patient does not have ability to operate study equipment, patient does not have a history of compliance to sending CareLink transmissions)
* Patients who have a reasonable probability of needing a device replacement during the study (approximately two months)
* Patients enrolled or planning to participate in a concurrent drug and/or device study during the course of this clinical trial
* Patient who are pregnant (all females of child-bearing potential must have a negative pregnancy test within 1 week of enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Adamson, MD, Principal Investigator — Oklahoma Cardiovascular Research
Locations (3):
- United States (3):
  - Ohio State University, Columbus, Ohio
  - Oklahoma Cardiovascular Research, Oklahoma City, Oklahoma
  - Sentara Cardiovascular, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Diuretic Adjustment
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 21
New York Heart Association Classification [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification classifies the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity.
  Class I: Cardiac disease, but no symptoms and no limitation in ordinary physical activity, Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III: Marked limitation in activity due to symptoms Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    Class I | 4
    Class II | 12
    Class III | 5
    Class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Characterize the Technical Feasibility of the Network Based IPC System
Description: The proportion of study days a PtIS is based on the subjects' daily pressure state
Time Frame: Baseline through Completion/Exit (an average of 3 months)
Population: The analysis population is the total number of study participants. For each study subject, the number of days in which the IPC system delivered a patient instruction set based on the subject's pressure state as measured by the Chronicle ICD/IHM pressure sensor.
Measure: Mean (95% Confidence Interval); unit: percentage of days
Units Other Than Participants: Days
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
Number analyzed (Days) | 1586
percentage of days | 72 [65 to 78]
Statistical Analysis 1: Comparison: Daily Diuretic Adjustment; Test type: Other — There was no specific hypothesis tested. The method of Rao and Scott for clustered binary data was used to construct a point estimate and 95% confidence interval for the number of days during the follow-up period across all subjects in which the patient instruction set was based on the subject's pressure state as measured by the Chronicle IHM/ICD system; Rao-Scott estimator for clustered data = 72, 95% CI 2-sided [65 to 78]

2. Secondary Outcome: Characterize the Rate of IPC Setup System Changes
Description: The frequency of changes in the IPC setup during the study (an average of 3-months).
Time Frame: Baseline through Completion/Exit (an average of 3-months)
Population: The analysis population is the total number of study participants. For each study subject, the number of changes to the IPC setup were obtained
Measure: Number (95% Confidence Interval); unit: changes per day
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
changes per day | 0.2 [0.1 to 0.4]

3. Secondary Outcome: Quantify Subject Compliance to Daily PtIS
Description: The proporition of IPC days study subjects indicated they complied with their PtIS.
Time Frame: Baseline through Completion/Exit (on average 3-months)
Population: The analysis population is the total number of study participants. For each study subject, the number of days in which the subject indicated that they followed their PtIS
Measure: Number (95% Confidence Interval); unit: proportion of compliant days
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
proportion of compliant days | 0.994 [0.988 to 1.000]

4. Secondary Outcome: Estimate Changes in Clinical Markers of Heart Failure and Kidney Function
Description: Changes in brain natriuretic peptide from baseline to study exit (an average of 3-months).
Time Frame: Baseline through Completion/Exit (an average of 3-months)
Population: Subjects with brain natriuretic peptide values at baseline and study completion (3-month visit) visits
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
pg/dL | -44.4 (388.8)

5. Secondary Outcome: Summarize Adverse Events
Description: All serious adverse events, cardiovascular adverse events, and event related to the IPC system will be documented and summarized.
Time Frame: Baseline through Completion/Exit (an average of 3-months)
Population: All 21 subjects participating in the IPC study
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
Participants
  Serious Adverse Event: Yes | 2
  Serious Adverse Event: No | 19
  IPC Related Adverse Events: Yes | 0
  IPC Related Adverse Events: No | 21
  PtIS Related Adverse Events: Yes | 0
  PtIS Related Adverse Events: No | 21
  Heart Failure Related Adverse Event: Yes | 2
  Heart Failure Related Adverse Event: No | 19
  Cardiovascular Related Adverse Event: Yes | 3
  Cardiovascular Related Adverse Event: No | 18

6. Secondary Outcome: Estimate Changes in Clinical Markers of Heart Failure and Kidney Function
Description: Changes in estimated glomular filtration rate from baseline to study exit (an average of 3-months).
Time Frame: Baseline through Completion/Exit (an average of 3-months)
Population: Subjects with lestimated glomular filtration rate values available at the baseline and study exit (3-month) visit.
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
mL/min per 1.73 m^2 | 0 (14.2)

7. Secondary Outcome: Estimate Changes in Clinical Markers of Heart Failure and Kidney Function
Description: Changes in blood urea nitrogen from baseline to study exit (an average of 3-months).
Time Frame: Baseline through Completion/Exit (an average of 3-months)
Population: Subjects with blood urea nitrogen values at both the baseline and study exit visits
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Daily Diuretic Adjustment
Number analyzed (Participants) | 21
mg/dL | 1 (6.2)

ADVERSE EVENTS:
Time Frame: All serious adverse events, cardiovascular related adverse events, and events related to the IPC system were captured from study enrollment through the study exit (approximately 60 days post-enrollment)
Arm/Group | Daily Diuretic Adjustment
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 4/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Diuretic Adjustment (N=21)
Cardiac Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Diuretic Adjustment (N=21)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The IPC study was a research feasibility study and was not powered to test any specific stastistical hypotheses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No